CLINICAL TRIAL: NCT00191854
Title: Randomized Phase II Study of Biweekly Gemcitabine-Paclitaxel, Biweekly Gemcitabine-Carboplatin and Biweekly Gemcitabine-Cisplatin as First-Line Treatment in Metastatic Breast Cancer After Anthracycline Failure
Brief Title: Gemcitabine Combinations in Metastatic Breast Cancer (MBC), 1st Line
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7451; B9E-AA-S355 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-08-31 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gemcitabine + Paclitaxel (Experimental): gemcitabine: 2500 milligrams per square meter (mg/m2), intravenous (IV), every 14 days x 8 cycles.
  paclitaxel: 150 mg/m2, IV, every 14 days x 8 cycles.
  Interventions: Drug: gemcitabine; Drug: paclitaxel
- Gemcitabine + Carboplatin (Experimental): gemcitabine: 2500 milligrams per square meter (mg/m2), intravenous (IV), every 14 days x 8 cycles.
  carboplatin: Area Under the Curve (AUC) 2.5, IV, every 14 days x 8 cycles.
  Interventions: Drug: gemcitabine; Drug: carboplatin
- Gemcitabine + Cisplatin (Experimental): gemcitabine: 2500 milligrams per square meter (mg/m2), intravenous (IV), every 14 days x 8 cycles.
  cisplatin: 50 mg/m2, IV, every 14 days x 8 cycles
  Interventions: Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: gemcitabine — 2500 milligrams per square meter (mg/m2), intravenous (IV), every 14 days x 8 cycles
  Other Names: LY188011; Gemzar
Drug: paclitaxel — 150 mg/m2, IV, every 14 days x 8 cycles
  Arms: Gemcitabine + Paclitaxel
Drug: carboplatin — Area Under the Curve (AUC) 2.5, IV, every 14 days x 8 cycles
  Arms: Gemcitabine + Carboplatin
Drug: cisplatin — 50 mg/m2, IV, every 14 days x 8 cycles
  Arms: Gemcitabine + Cisplatin

SUMMARY:
The gemcitabine-paclitaxel and gemcitabine-platinum combinations have shown promise in the treatments of MBC; however, the optimal dosing schedules for these combinations have not yet been determined. The primary objective of this study is to compare the response rates of the gemcitabine-paclitaxel, gemcitabine-carboplatin, and gemcitabine-cisplatin combinations when administered on a biweekly schedule in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histological or cytological proven diagnosis of breast cancer
* Stage IV disease
* Performance Status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Scale
* Patients had to have previously received anthracycline based regimens as a adjuvant therapy or neo-adjuvant chemotherapy and then progressed and developed metastatic disease
* Adequate organ function

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Previous radiation therapy is allowed but must not have included whole pelvis radiation
* Known or suspected brain metastasis. Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy and immunotherapy (including trastuzumab (Herceptin))
* Peripheral neuropathy of Common Toxicity Criteria (CTC) Grade greater than 1. History of significant neurological or mental disorder, including seizures or dementia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2005-03; Primary Completion 2008-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Monday-Friday 9:00 AM to 5:00 PM Est Time (UTC/GMT - 5 hours), Study Director — Eli Lilly and Company
Locations (18):
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santo André
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- China (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludhiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villahermosa
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin
Started | 49 | 47 | 51
Received at Least One Dose of Study Drug | 49 | 47 | 50 (Screen failure: discontinued prior to receiving study drug.)
Completed | 12 | 17 | 12
Not Completed | 37 | 30 | 39
Not completed — Death | 26 | 23 | 29
Not completed — Lost to Follow-up | 7 | 5 | 5
Not completed — Withdrawal by Subject | 4 | 2 | 3
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Screen Failure | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 49 | 47 | 51 | 147
Age Continuous [Mean (Standard Deviation); unit: years] | 49.8 (8.8) | 46.0 (6.9) | 49.2 (10.3) | 48.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 51 | 147
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 1 | 2 | 3 | 6
  Brazil | 5 | 5 | 4 | 14
  Turkey | 5 | 2 | 4 | 11
  China | 25 | 25 | 26 | 76
  Korea, Republic of | 5 | 5 | 6 | 16
  India | 8 | 8 | 8 | 24
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 22 | 29 | 26 | 77
    1 - Ambulatory, Restricted Strenuous Activity | 27 | 18 | 24 | 69
    Missing Data | 0 | 0 | 1 | 1
Menopausal Status [Number; unit: participants]
  Pre-Menopausal | 11 | 16 | 13 | 40
  Peri Menopausal | 4 | 4 | 4 | 12
  Post Menopausal | 34 | 26 | 33 | 93
  Missing Data | 0 | 1 | 1 | 2
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma | 1 | 2 | 2 | 5
  Carcinoma, Infiltrating Ductal | 42 | 40 | 45 | 127
  Carcinoma, Infiltrating Lobular | 6 | 4 | 2 | 12
  Carcinoma, Undifferentiated | 0 | 1 | 0 | 1
  Comedocarcinoma | 0 | 0 | 1 | 1
  Missing Data | 0 | 0 | 1 | 1
Race/Ethnicity [Number; unit: participants]
  African | 1 | 0 | 1 | 2
  Caucasian | 8 | 6 | 7 | 21
  East Asian | 30 | 30 | 32 | 92
  Hispanic | 2 | 3 | 3 | 8
  West Asian (West Indian) | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (tumor assessments were performed every 4 cycles during study therapy, or 3 months during post-therapy until disease progression, death or up to 24 months after randomization)
Population: Number of all randomized participants.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49 | 47 | 51
participants
  Complete Response (CR) | 1 | 0 | 1
  Partial Response (PR) | 12 | 8 | 7
  Stable Disease (SD) | 17 | 25 | 29
  Progressive Disease (PD) | 14 | 11 | 11
  Early Death from Other Causes | 1 | 2 | 0
  Unknown | 4 | 1 | 3

2. Secondary Outcome: Number of Participants With a Time to Treatment Failure (TTTF) Event
Description: TTTF event was defined as documented disease progression, death on study, start of non-protocol-specified anticancer therapy, or therapy discontinuation due to toxicity. TTTF for patients who were still participating in study without treatment failure at time of analysis were treated as censored at date of last tumor assessment. TTTF for patients who had discontinued from therapy for reasons other than toxicity and who did not experience treatment failure prior to therapy discontinuation were treated as censored on day of study discontinuation.
Time Frame: randomization to date of documented disease progression, death on study, start of non-protocol-specified anticancer therapy, or therapy discontinuation due to toxicity, whichever occurred first (up to 6 months)
Population: Number of randomized patients. Censored patients: Gemcitabine + Paclitaxel = 34; Gemcitabine + Carboplatin = 26; Gemcitabine + Cisplatin = 30.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49 | 47 | 51
participants | 15 | 21 | 21

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomizaton to the date of documented disease progression or death on study, whichever occurred first. PFS for participants who discontinued from the study or who had not progressed at the time of analysis were treated as censored at the date of the last tumor assessment.
Time Frame: baseline to measured progressive disease or death (tumor assessments were performed every 4 cycles during study therapy, or 3 months during post-therapy until disease progression, death, or up to 24 months after randomization)
Population: Number of randomized patients. Censored patients: Gemcitabine + Paclitaxel = 20; Gemcitabine + Carboplatin = 18; Gemcitabine + Cisplatin = 28.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49 | 47 | 51
months | 4.8 [4.2 to 7.0] | 4.3 [3.7 to 5.9] | 4.8 [3.7 to 8.1]

4. Secondary Outcome: Duration of Response
Description: Duration of response was measured from time of first documentation of complete response (disappearance of all target lesions) or partial response (30% decrease in sum of longest diameter of target lesions), until date of PFS. Duration of response was censored on day of last tumor assessment for patients who had not progressed or who had discontinued study at time of analysis, and for cases where investigator determined patient had progressive disease and discontinued study therapy and/or started a new, non-protocol-specified anti-cancer therapy before documented disease progression.
Time Frame: time of response to progressive disease or death (tumor assessments were performed every 4 cycles during study therapy, or 3 months during post-therapy until disease progression, death, or up to 24 months after randomization)
Population: Randomized patients who had either a complete response or partial response. Censored patients: Gemcitabine + Paclitaxel = 4; Gemcitabine + Carboplatin = 4; Gemcitabine + Cisplatin = 14.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 13 | 8 | 8
months | 5.8 [4.9 to 8.1] | 3.2 [1.9 to 5.0] | 5.1 [2.9 to 5.1]

5. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from the date of randomization to date of death due to any cause. Survival time is censored at the date of last contact for patients who are still alive or lost to follow-up.
Time Frame: baseline to date of death from any cause (up to 34 months)
Population: Number of randomized patients. Censored patients: Gemcitabine + Paclitaxel = 23; Gemcitabine + Carboplatin = 24; Gemcitabine + Cisplatin = 22.
Measure: Median (Full Range); unit: months
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49 | 47 | 51
months | 15.5 [0.361 to 33.84] | 22.8 [1.413 to 26.12] | 20.1 [1.413 to 27.83]

ADVERSE EVENTS:
Description: Safety analyses were performed on all enrolled patients who received at least one dose of study therapy. All enrolled patients, except for one patient in Gemcitabine + Cisplatin Arm, received at least one dose of study therapy and qualified for safety analyses. The one patient was a screen failure and was discontinued before receiving study drug.
Arm/Group | Gemcitabine + Paclitaxel | Gemcitabine + Carboplatin | Gemcitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 5/49 | 3/47 | 0/50
Other Adverse Events (participants affected / at risk) | 48/49 | 46/47 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Paclitaxel (N=49) | Gemcitabine + Carboplatin (N=47) | Gemcitabine + Cisplatin (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Paclitaxel (N=49) | Gemcitabine + Carboplatin (N=47) | Gemcitabine + Cisplatin (N=50)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (11) | 9 (13) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 8 (12) | 2 (2) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 9 (17) | 10 (11) | 6 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 5 (7) | 3 (7)
Palpitations (Cardiac disorders) | 0 (0) | 3 (4) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (9) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (11) | 10 (17) | 9 (21)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 5 (5) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (5)
Nausea (Gastrointestinal disorders) | 19 (53) | 25 (61) | 39 (161)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 12 (21) | 22 (57) | 31 (127)
Asthenia (General disorders) | 2 (9) | 3 (5) | 6 (12)
Fatigue (General disorders) | 18 (32) | 17 (36) | 15 (29)
Mucosal inflammation (General disorders) | 4 (6) | 0 (0) | 1 (1)
Oedema (General disorders) | 5 (6) | 3 (5) | 2 (2)
Pyrexia (General disorders) | 8 (12) | 8 (9) | 6 (11)
Infection (Infections and infestations) | 3 (7) | 2 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 18 (27) | 20 (22) | 8 (13)
Aspartate aminotransferase increased (Investigations) | 14 (20) | 14 (18) | 6 (9)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 5 (9) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 4 (5) | 2 (2)
Haemoglobin decreased (Investigations) | 15 (31) | 18 (20) | 18 (27)
Neutrophil count decreased (Investigations) | 22 (45) | 14 (28) | 21 (40)
Platelet count decreased (Investigations) | 7 (9) | 18 (25) | 7 (13)
White blood cell count decreased (Investigations) | 17 (41) | 13 (26) | 13 (28)
Anorexia (Metabolism and nutrition disorders) | 11 (22) | 15 (28) | 8 (18)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (5)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (8) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (22) | 4 (6) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (46) | 5 (16) | 7 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 6 (9) | 5 (8) | 5 (9)
Hypoaesthesia (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (16) | 3 (7) | 4 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (5) | 1 (1) | 4 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 9 (9) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (11) | 6 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 25 (26) | 16 (16) | 22 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (8) | 10 (11) | 8 (11)
Hypertension (Vascular disorders) | 4 (4) | 3 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days